CLINICAL TRIAL: NCT05701696
Title: Investigation of the Relationship Between Neuropathic Complaints and Central Sensitization in Patients With Fibromyalgia
Brief Title: The Relationship Between Neuropathic Complaints and Central Sensitization in Fibromyalgia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 22/640
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-01

CONDITIONS: Central Sensitisation; Fibromyalgia; Neuropathic Pain
MeSH Terms: conditions — Fibromyalgia; Neuralgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with fibromyalgia: Patients diagnosed with FM according to ACR 2016 criteria
  Interventions: Diagnostic Test: Central sensitization inventory; Diagnostic Test: Widespread pain index; Diagnostic Test: Symptom severity scale; Other: Fibromyalgia impact questionnaire; Diagnostic Test: Hospital Anxiety and Depression Scale; Diagnostic Test: Self-Leeds Assessment of Neuropathic Symptoms and Signs

INTERVENTIONS:
Diagnostic Test: Central sensitization inventory — Standardized questionnaire to determine the level of central sensitization. Patients with a score of 40 and above are considered to have central sensitization.
  Other Names: CSI
Diagnostic Test: Widespread pain index — Total the number of painful body areas
  Other Names: WPI
Diagnostic Test: Symptom severity scale — The sum of the fatigue, waking unrefreshed and cognitive symptoms and the extent of somatic symptoms
  Other Names: SSS
Other: Fibromyalgia impact questionnaire — A tool to assess health status in fibromyalgia
  Other Names: FIQ
Diagnostic Test: Hospital Anxiety and Depression Scale — An instrument for detecting depression and anxiety
  Other Names: HADS
Diagnostic Test: Self-Leeds Assessment of Neuropathic Symptoms and Signs — An instrument used to identify pain of neuropathic origin
  Other Names: S-LANSS

SUMMARY:
Fibromyalgia (FM) is the prototype of a group of diseases known as central sensitivity syndromes, whose relationship with pain sensitization is well defined. Central sensitization (CS) is also one of the mechanisms involved in the pathophysiology of neuropathic pain. Neuropathic pain, which is a common complaint in FM patients, is likely to be one of the clinical manifestations of central sensitization. Therefore, in this study, it was aimed to investigate the relationship between CS and neuropathic pain.

DETAILED DESCRIPTION:
The term central sensitization (CS) was first used by Wolf in 1988 and explained as an increase in pain sensitivity with the amplification of neuron-derived signals in the central nervous system. Fibromyalgia (FM) is a disease characterized by chronic widespread pain and its etiology and pathophysiology are still unknown. It is considered to be the main member of the CS related disease group known as central sensitivity syndromes with impaired pain regulation. In various studies, hyperalgesia and allodynia, which are accepted as objective findings of CS in pain sensitization. In addition to widespread body pain, neuropathic pain is one of the common symptoms in FM, and various studies have shown a significant increase in neuropathic pain in FM patients compared to healthy controls. It is known that CS is one of the basic mechanisms in the etiopathogenesis of neuropathic pain as well as its role in FM. In a study of FM patients, painDETECT and S-LANSS scores were found to be correlated with CSI scores, and the authors emphasized the relationship between pain sensitization and neuropathic complaints in these patients. CS seems likely to be one of the neuropathic pain mechanisms in FM patients, and the available data seem insufficient to draw a definitive conclusion. From this point of view, in this study, it was aimed to investigate the relationship between the presence and severity of CS and the neuropathic pain component of the disease in patients with FM.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosing fibromyalgia according to ACR 2016 criteria
* Between the ages of 18-65
* Agree to participate in the study

Exclusion Criteria:

* History of concomitant systemic inflammatory disease, active infection and malignancy
* Refusing to participate in the study
* Polyneuropathy, entrapment neuropathy, and radiculopathy are other diagnosed sources of neuropathic pain.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Fibromyalgia patients
Sampling Method: Non-Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
CSI | 1 year
  Standardized questionnaire to determine the level of central sensitization. Patients with a score of 40 and above are considered to have central sensitization.
S-LANSS | 1 year
  Questionnaire used to investigate the neuropathic character of pain. A score ≥12 points suggests the presence of pain of neuropathic origin

SECONDARY OUTCOMES:
Visual analog scale ( VAS) pain | 1 year
  Pain rating scale. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
Fibromyalgia impact scale | 1 year
  The questionnaire was developed to determine the degree of being affected by the disease in patients with a diagnosis of fibromyalgia.The scale consists of 10 parts in total, and the first part is a Likert scale containing 11 questions. High scores indicate that the patient is overly affected.
Symptom severity scale | 1 year
  The SS scale quantifies symptom severity on a 0-12 scale by scoring problems with fatigue, cognitive dysfunction and unrefreshed sleep over the past week. SSI ≥ 5 favors fibromyalgia.
Widespread pain index | 1 year
  In this scale, the areas with pain in the last 7 days are marked from a total of 5 regions, including the right and left upper region, the right and left lower region, and the axial region. The total score is between 0-19, and YAS ≥ 7 points is significant for the diagnosis of fibromyalgia.
HADS | 1 year
  The scale consists of 14 questions, 7 of which are anxiety and 7 are depression.More than 10 points for anxiety and 7 points for depression are considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Feyza Nur Yücel, MD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woolf CJ, Thompson SW, King AE. Prolonged primary afferent induced alterations in dorsal horn neurones, an intracellular analysis in vivo and in vitro. J Physiol (Paris). 1988-1989;83(3):255-66. PMID 3272296
- [Background] Bhargava J, Goldin J. Fibromyalgia. 2025 Jan 31. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK540974/ PMID 31082018
- [Background] Pomares FB, Funck T, Feier NA, Roy S, Daigle-Martel A, Ceko M, Narayanan S, Araujo D, Thiel A, Stikov N, Fitzcharles MA, Schweinhardt P. Histological Underpinnings of Grey Matter Changes in Fibromyalgia Investigated Using Multimodal Brain Imaging. J Neurosci. 2017 Feb 1;37(5):1090-1101. doi: 10.1523/JNEUROSCI.2619-16.2016. Epub 2016 Dec 16. PMID 27986927
- [Background] Martinez-Lavin M. Fibromyalgia in women: somatisation or stress-evoked, sex-dimorphic neuropathic pain? Clin Exp Rheumatol. 2021 Mar-Apr;39(2):422-425. doi: 10.55563/clinexprheumatol/0c7d6v. Epub 2020 Sep 16. PMID 32940205
- [Background] Ubeda-D'Ocasar E, Valera-Calero JA, Gallego-Sendarrubias GM, Fernandez-de-Las-Penas C, Arias-Buria JL, Morales-Cabezas M, Arendt-Nielsen L, Cigaran-Mendez M. Association of Neuropathic Pain Symptoms with Sensitization Related Symptomatology in Women with Fibromyalgia. Biomedicines. 2022 Mar 6;10(3):612. doi: 10.3390/biomedicines10030612. PMID 35327414
- [Background] Bennett M. The LANSS Pain Scale: the Leeds assessment of neuropathic symptoms and signs. Pain. 2001 May;92(1-2):147-57. doi: 10.1016/s0304-3959(00)00482-6. PMID 11323136
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820